CLINICAL TRIAL: NCT04943458
Title: Application of Innovative Non-Invasive Neuroprotective Technology in Cardiac Surgery and Ophthalmology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Milda Svagzdiene (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Sponsor-Investigator, Milda Svagzdiene, dr, assoc. prof., Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: Nr.1
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Cognitive Disorder; Glaucoma
MeSH Terms: conditions — Postoperative Cognitive Complications; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiac surgery group
  Interventions: Other: Monitoring of cerebral autoregulation
- Glaucoma group
  Interventions: Other: Monitoring of cerebral autoregulation
- Control group
  Interventions: Other: Monitoring of cerebral autoregulation

INTERVENTIONS:
Other: Monitoring of cerebral autoregulation — Patients will be monitored for cerebral autoregulation using a Vittamed 505 monitor to identify the dynamics of the autoregulation index VRx (t). Intracranial pressure (ICP) will also be measured by non-invasive ultrasound using a robotic TCD device, Dolphin4D (Israel), which simultaneously records MCA blood flow in both hemispheres of the brain. APAs will be assessed using mathematical models.
  Other Names: Non invasive ICP monitoring

SUMMARY:
Postoperative cognitive dysfunction (POCD) and delirium (incidence up to 42 %) after cardiac surgery with cardiopulmonary bypass (CPB) are common postoperative complications that impair the patient's quality of life and increase the risk of death. Our previous studies confirm that postoperative POCD are associated with impaired cerebral autoregulation (CA) and momentary increased intracranial pressure (ICP) during surgery. The upper and lower limits of CA are individual and variable. In the elderly, CA is already partially impaired due to decreased cerebral vascular elasticity. What should be the optimal mean arterial pressure for each of these patients individually is not known. In order to individualize the boundaries of CA and prevent postoperative neurological complications, it would be ideal to objectify the condition of cerebral blood vessels. Direct studies of cerebrovascular and vascular status (CT angiography) are invasive and complex, and are therefore not routinely performed prior to cardiac surgery. However, cerebral blood flow and vascular condition can be assessed by retinal blood vessels, which can be considered as a direct biomarker of cerebrovascular disorders and can be visualized by ophthalmoscopy and objectively assessed by optical coherent tomography with angiography.

In this biomedical study, individual patient CA will be monitored in a non-invasive manner during cardiac surgery with CPB. These data would allow real-time adjustments to physiological parameters while keeping them within normal limits. This is expected to reduce the risk of CA impairment and reduce the incidence of neurological complications following such surgery.

Glaucoma is one of the leading causes of irreversible blindness in the world. As the population ages, the number of people with glaucoma increases as the prevalence of glaucoma increases with age. Recently, the influence of ICP on glaucoma optic neuropathy has been highlighted. It is thought that the pressure difference in the optic nerve area may be related to damage to the axons of the ganglion cells passing through the porous plate. Noninvasive ICP measurement is useful in explaining the pathophysiology of glaucoma, assessing translaminar pressure differentials, and seeking new guidelines for the treatment and prevention of glaucoma. Retinal blood flow, like cerebral blood flow, is autoregulated, autoregulation is maintained only within certain limits of perfusion pressure. Decreased ocular perfusion pressure impairs retinal autoregulation and may lead to the development or progression of glaucoma neuropathy. And the activity of neurons in the brain and retina causes local changes in blood circulation. Disruption of this neurovascular interaction during glaucoma neuropathy has not been adequately studied.The introduction of modern technologies into clinical practice enables the qualitative and quantitative assessment of autoregulatory disorders and the selection of optimal treatment.

ELIGIBILITY:
Inclusion Criteria:

I. Criteria for the inclusion of the CA monitoring method in cardiac surgery:

1. Age 18-90 years.
2. The patient, after reading the personal information form, confirms in writing his / her consent to participate in the study.
3. An AVJS operation is planned.
4. No ophthalmological or neurological disorders have been identified prior to surgery.

II. Criteria for the inclusion of the CA monitoring method in ophthalmology:

1. Age 18-90 years.
2. The patient, after reading the personal information form, confirms in writing his / her consent to participate in the study.
3. Patients with glaucoma changes in the optic disc and eye area shall be included in the study group.
4. The control group shall include volunteers who are free from glaucoma, acute or chronic uncompensated disease that may affect the results of the studies, and age and anthropometric data from other study groups.

Exclusion Criteria:

1. No written consent of a person to participate in a biomedical research has been obtained;
2. Persons under 18 years of age.
3. A woman who may become pregnant, be pregnant or breastfeeding.
4. The patient is allergic or sensitive to local anesthetics.
5. Patients with an eye disease that may distort the results of the test, if so decided by the researcher.
6. The patient had an orbital or eye injury.
7. Has an acute or chronic but currently exacerbated respiratory disease.
8. Patients with uncompensated cardiovascular diseases (II-III AV block or cardiogenic shock).
9. Diabetes mellitus treated with more than one hypoglycaemic agent and / or insulin injections.
10. Cognitive impairment diagnosed before surgery
11. History of neurological diseases
12. It is not possible to perform a qualitative neuropsychological examination due to other reasons (hearing, vision, etc. disorders)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients treated at the Clinic of Eye Diseases, Hospital of Lithuanian UHS and patients undergoing elective cardiac surgery (coronary artery bypass graft surgery) at the Clinic of Cardiovascular and Thoracic Surgery, Hospital of Lithuanian UHS.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Impaired cerebral autoregulation and glaucoma neuropathy | 1 days
  Duration of the longest episode of CA disorder (threshold VRx> 0, threshold VRx> 0.2, threshold VRx> 0.4) showing impaired CA and the changes in vascular density ( %) of OCT-A macular temporal sector assessing the course of glaucoma neuropathy.

SECONDARY OUTCOMES:
POCD and glaucoma neuropathy | 5 days up to 1 month
  . Postoperative cognitive impairment. Changes in vascular density (%) of the lower temporal sector of the OCT-A optic nerve disc for monitoring structural changes in glaucoma neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Milda Svagzdiene, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No